CLINICAL TRIAL: NCT00552500
Title: Effects of Atypical Antipsychotic and Valproate Combination Therapy on Glucose and Lipid Metabolism in Schizophrenia
Acronym: DepIVGTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NARSAD 43625; NARSAD; NCT00161512 (obsolete NCT alias)
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Insulin Resistance; Body Composition
MeSH Terms: conditions — Insulin Resistance | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Schizophrenics (Active Comparator): i) meets DSM-IV criteria for schizophrenia, any type, treated with atypical or high potency typical neuroleptics for at least 3 months; ii) aged 18 to 60 years; iii) able to give informed consent; iv) no antipsychotic medication changes for 3 months, and no other medication changes for 2 weeks prior to Baseline Evaluations.
  Interventions: Drug: Depakote (valproate)

INTERVENTIONS:
Drug: Depakote (valproate) — 500 mg -2000 mg QD based on individual tolerance and VPA levels

SUMMARY:
This project aims to a) evaluate the effects of haloperidol, olanzapine, and risperidone in combination with valproate on insulin secretion and insulin actions, b) evaluate medication effects on abdominal fat, total body fat and total fat-free mass, and c) evaluate treatment effects on glucose tolerance, lipid profiles, and plasma levels of leptin, adiponectin, ghrelin and C-reactive protein. Hypotheses will be evaluated by measuring 1) insulin action and secretion using frequently sampled intravenous glucose tolerance tests, 2) body composition using dual energy x-ray absorptiometry, magnetic resonance scans, and anthropomorphic measurements, and 3) changes in hormone levels and lipid profiles. The aims will be addressed in non-diabetic schizophrenia patients chronically treated with haloperidol, olanzapine or risperidone who will have valproate added to their treatment. Relevant data is critically needed to target basic research, identify long-term cardiovascular risks, and plan therapeutic interventions.

DETAILED DESCRIPTION:
Schizophrenia is associated with increased rates of obesity, hyperglycemia, dyslipidemia and type 2 diabetes mellitus, causing increased morbidity and mortality due to acute (e.g., diabetic ketoacidosis) and long-term (e.g., vascular disease) complications. The association of type 2 diabetes and hyperglycemia with schizophrenia was first noted prior to the introduction of antipsychotic medications. However, additional glucoregulatory abnormalities, dyslipidemia, and increased adiposity have all been associated with antipsychotics. Risperidone and olanzapine are the most prescribed antipsychotics for schizophrenia in the U.S. In addition, schizophrenia patients in clinical practice are commonly treated with multi-class polypharmacy, with 35% of atypical antipsychotic prescriptions accompanied by co-prescription of valproate. This combination continues to increase in popularity, despite reports that the addition of valproate may further disturb glucose and lipid metabolism and weight regulation. While sensitive and validated measures of glucose and lipid metabolism and weight regulation are available, very few studies have addressed the metabolic consequences of this common type of polypharmacy.

This project aims to a) evaluate the effects of haloperidol, olanzapine, and risperidone in combination with valproate on insulin secretion and insulin actions, b) evaluate medication effects on abdominal fat, total body fat and total fat-free mass, and c) evaluate treatment effects on glucose tolerance, lipid profiles, and plasma levels of leptin, adiponectin, ghrelin and C-reactive protein. Hypotheses will be evaluated by measuring 1) insulin action and secretion using frequently sampled intravenous glucose tolerance tests, 2) body composition using dual energy x-ray absorptiometry, magnetic resonance scans, and anthropomorphic measurements, and 3) changes in hormone levels and lipid profiles. The aims will be addressed in non-diabetic schizophrenia patients chronically treated with haloperidol, olanzapine or risperidone who will have valproate added to their treatment. Relevant data is critically needed to target basic research, identify long-term cardiovascular risks, and plan therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia, any type, treated with atypical or high potency typical neuroleptics for at least 3 months
* Aged 18 to 60 years
* Able to give informed consent
* No antipsychotic medication changes for 3 months, and no other medication changes for 2 weeks prior to Baseline Evaluations.

Exclusion Criteria:

* Meets DSM-IV criteria for the diagnoses of substance abuse or dependence within the past 6 months
* Involuntary legal status (as per Missouri law)
* The presence of any serious medical disorder that may (as confirmed by peer-reviewed literature) confound the assessment of symptoms, relevant biologic measures or diagnosis. The following conditions are currently identified:

  * Type 1 diabetes mellitus or symptomatic type 2 diabetes mellitus
  * Any intra-abdominal or intrathoracic surgery or limb amputation within the prior 6 months
  * Any diagnosed cardiac condition causing documented hemodynamic compromise
  * Any diagnosed respiratory condition causing documented or clinically recognized hypoxia
  * Pregnancy or high dose estrogens, fever, narcotic therapy, acute sedative hypnotic withdrawal, corticosteroid or spironolactone therapy, dehydration, epilepsy, endocrine disease, high-dose benzodiazepine therapy (> 25 mg/day of diazepam), or any medical condition known to interfere with glucose utilization
* Meets DSM-IV criteria for Mental Retardation (mild or worse).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-02 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Hypotheses will be evaluated by measuring insulin action and secretion using frequently sampled intravenous glucose tolerance tests | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Haupt, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States